CLINICAL TRIAL: NCT07193875
Title: Safety, Tolerability, and Efficacy of Efavirenz (EFV) Intensification on HIV-1 Reservoir Reduction
Brief Title: Efavirenz (EFV) Intensification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Rachel Presti, Associate Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202210153
Record Dates: First submitted 2025-09-16; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2023-01

CONDITIONS: HIV
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Intervention Model Description: Each participant will be their own control for size of latent reservoir. We will compare each person's reservoir before and after addition of Efavirenz.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Efavirenz intensification (Other): There is only one arm in this study
  Interventions: Drug: Efavirenz 600mg

INTERVENTIONS:
Drug: Efavirenz 600mg — Take One pill daily for 6 months in addition to baseline combination antiretroviral therapy regimen

SUMMARY:
The goal of this clinical trial is to see if Efavirenz (EFV) intensification to a baseline combination antiretroviral regimen (cART) can help reduce the size of the latent reservoir in people living with HIV (PLWH). The main questions this study aims to address are:

1. is the addition of EFV to a cART regimen safe and well tolerated?
2. Is there a reduction in the blood and tissue HIV reservoir after intensification?

Researchers will compare each participants reservoir size prior to and post EFV intensification.

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of efavirenz (EFV) intensification on the HIV-1 reservoir. Participants with well controlled HIV, specifically with a HIV VL <500 for at least 48 weeks will be eligible. Prior to enrollment, we will prescreen individuals to ensure they do not have a polymorphism in CY450 which results in rapid metabolism of the study drug efavirenz. Leukapheresis and lymph node (LN) fine needle aspirates will be collected at baseline. Participants eligible to participate will begin taking Efavirenz in addition to their baseline combination antiretroviral therapy. Blood samples (120ml) will be collected twice at day 30 and day 90 for cell associated HIV RNA and HIV DNA assessments. Follow-up LN aspirates and follow-up Leukapheresis will be collected at completion of study, between day 150-180, based on scheduling. At day 90 pharmacokinetic (PK) evaluation of EFV will take place to ensure therapeutic levels of Efavirenz. At the completion of the 180 day course of efavirenz, participants will stop efavirenz but continue their baseline HIV regimen. CD4, HIV VL and monitoring chemistries will be performed at visits on day 30, day 90 and day 150-180.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Diagnosis of HIV
3. Documentation of at least two historical HIV-1 RNA measurements <500 copies/mL while on ART obtained by standard assay.
4. No known non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance mutations.
5. Currently on a stable regimen including an integrase strand transfer inhibitor (INSTI) and two nucleoside reverse transcriptase inhibitors (NRTI). Receiving the current regimen for at least 90 days prior to study entry with no intention to change for the duration of the study.

Exclusion Criteria:

1. Untreated depression, defined as a PHQ-9 > 15 at time of enrollment
2. Known prior NNRTI resistance, or INSTI resistance.
3. Cytochrome 450 polymorphism resulting in rapid or delayed metabolism of Efavirenz
4. Not currently on a PI based regimen.
5. Does not have an immunocompromising medical condition. (ie malignancies particularly leukemia, lymphoma, use of immunosuppressive or antineoplastic drugs or X-ray treatment).
6. Chronic, acute, or recurrent infections that are current and serious, in the opinion of the site investigator.
7. Breastfeeding patients as well as those whom are pregnant or plan to become pregnant during period of the study.
8. Those with active Hepatitis C or Hepatitis B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Safety of Efavirenz intensification on a baseline cART regimen | 3 months post completion of trial
  Safety of Efavirenz intensification on a baseline cART regimen
  The safety will be addressed both with laboratory tests (CBC, CMP, CD4, HIV VL) performed monthly, and PHQ9 surveys (for the rare reported adverse effect of worsening depression with Efavirenz) in addition to asking patients more subjective questions of how they are feeling and tolerating the medications and self reporting of (rash, pruritis, mood changes, nausea, vomiting or new abnormal symptoms).

SECONDARY OUTCOMES:
Size of the latent reservoir | within 2 years post study completion
  Size of intact provirus pre and post Efavirenz intensification as measured by IPDA

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
we plan to analyze the data and publish this in an accessible manuscript to the public
Supporting Information: CSR
Time Frame: within 3 years of study completion
Access Criteria: depends on the journal the study results are published in

REFERENCES:
- [Background] Barnthouse LW. Issues in ecological risk assessment: the CRAM perspective. Risk Anal. 1994 Jun;14(3):251-6. doi: 10.1111/j.1539-6924.1994.tb00239.x. PMID 8029496